CLINICAL TRIAL: NCT02367248
Title: Safety and Effectiveness Study of Deferoxamine and Xingnaojing Injection in Intracerebral Hemorrhage
Brief Title: Deferoxamine and Xingnaojing Injection Treatment in Intracerebral Hemorrhage
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Collaborators: Beijing Tiantan Hospital (Other); Peking University First Hospital (Other); People's Hospital of Beijing Daxing District (Other); Beijing Haidian Hospital (Other); The 263 Hospital of PLA (Unknown); Beijing Aerospace General Hospital (Other); Peking University Third Hospital (Other); Beijing Pinggu District Hospital (Other); Beijing Shuyi Hospital (Other); General Hospital of Beijing PLA Military Region (Other); Beijing Luhe Hospital (Other); Beijing Fangshan District Liangxiang Hospital (Other); Beijing Neurosurgical Institute (Other); Beijing Jishuitan Hospital (Other); Beijing Ditan Hospital (Other); Beijing Youyi Hospital (Unknown); Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other); Peking University People's Hospital (Other); The Second Artillery General Hospital (Other); Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Maolin He, director of the Neurology department, Beijing Shijitan Hospital, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MHe
Record Dates: First submitted 2015-02-13; First posted 2015-02-20 (Estimated); Last update posted 2015-05-18 (Estimated); Status verified 2015-05

CONDITIONS: Intracerebral Hemorrhage
Keywords: Brain hemorrhage; Cerebral Hemorrhage; Deferoxamine; Xingnaojing injection; Hematoma edema
MeSH Terms: conditions — Cerebral Hemorrhage; Intracranial Hemorrhages | interventions — Deferoxamine; xingnaojing; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Deferoxamine (Active Comparator): Deferoxamine mesylate supplied in vials containing 500 mg of sterile, lyophilized, powdered deferoxamine mesylate. The drug will be reconstituted for injection, by dissolving in 20 ml of sterile water.
  Interventions: Drug: deferoxamine
- Xingnaojing injection (Active Comparator): Xingnaojing injection supplied in vials containing 20 ml liquid xingnaojing.
  Interventions: Drug: Xingnaojing injection
- Normal Saline (Placebo Comparator): 0.9% sodium chloride
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: deferoxamine — Deferoxamine mesylate(40 mg/kg/day up to a maximum daily dose of 6000 mg/day) given by a continuous IV infusion for 5 consecutive days beginning within 12 hours of ICH symptom onset.
  Other Names: Deferoxamine Mesylate
  Arms: Deferoxamine
Drug: Xingnaojing injection — Xingnaojing injection (20 ml/day) given by a continuous IV infusion for 5 consecutive days beginning within 12 hours of ICH symptom onset.
  Arms: Xingnaojing injection
Drug: Normal saline — This is a placebo. Normal saline will be given by a continuous IV infusion for 5 consecutive days beginning within 12 hours of ICH symptom onset.
  Other Names: 0.90% Sodium Chloride Solution
  Arms: Normal Saline

SUMMARY:
The main purpose of this study is to determine whether deferoxamine and xingnaojing injection is effective and safe as a treatment for intracerebral hemorrhage.

DETAILED DESCRIPTION:
Research shows that more than 1/3 of patients with acute cerebral hemorrhage in the first 24 hours will be expanding hematoma. The treatment of acute cerebral hemorrhage has two main targets: prevention of hematoma enlargement in primary brain damage; Reduce hematoma secondary brain damage caused by blood toxicity degradation products. At present, the curative effect of drug treatment of acute cerebral hemorrhage remains limited, using drug therapy to treat hematoma caused by blood toxicity degradation products secondary brain damage, is one of the main current international research direction and hotspot. Recent studies have found that iron overload in cells in acute cerebral hemorrhage stove weeks edema secondary lesion plays a very important role. Acute cerebral hemorrhage animal model research and small sample clinical study has shown that the iron chelator deferoxamine has good curative effect and security. Currently ongoing international HI-DEF test plans to assess the efficacy and safety of high-dose deferoxamine treatment within 24 h of patients with acute cerebral hemorrhage.

Basic research shows Xingnaojing injection can inhibit inflammatory reaction, scavenging free radicals, relieve acute cerebral hemorrhage hematoma surrounding edema and has a variety of brain protection mechanism. The current study builds on these results to assess the potential utility of deferoxamine and Xingnaojing injection as a therapeutic intervention in ICH.

This is a prospective, multi-center, double-blind, randomized, placebo-armed clinical study to test the safety and effectiveness of deferoxamine and Xingnaojing injection treatment in intracerebral hemorrhage. The investigators will randomize 180 subjects with ICH equally (1:1:1) to either DFO at 40mg/kg/day (up to a maximum daily dose of 6000 mg/day), or Xingnaojing injection, or saline placebo, given by continuous IV infusion for 5 consecutive days. Treatment will be initiated within 12 hours after ICH symptom onset.

The main objectives are:

1. Examining the effects of DFO and Xingnaojing injection on peri-hematoma edema (PHE) volume progression between baseline and post-treatment CT/MRI scans and the residual cavity volume at 90 days.
2. Obtaining data on the National Institute of Health Stroke Scale (NIHSS) to explore the effects of treatment on neurological functions.
3. Examining the effects of DFO and Xingnaojing injection on biomarkers of acute cerebral hemorrhage such as ferritin, interleukin - 6, matrix metalloproteinase 9, tumor necrosis factor alpha and so on.
4. Study the traditional Chinese medicine(TCM)curative effect evaluation of the roles of different treatment methods on secondary damage after ICH.

Secondary and exploratory objectives include:

1. Exploring whether the effect of DFO on outcome is dependent on initial ICH volume, after adjusting for other prognostic variables, to determine if specific limits for ICH volume should be specified as exclusion/inclusion criteria for future studies.
2. Exploring the differences between early (≤12h) and late (>12-24h) OTT windows in DFO treatment effect on functional outcome.

Exploratory study shows that iron chelator deferoxamine is effective and safe in the treatment of acute cerebral hemorrhage. We choose within 12 hours as the treatment time window, different from within 24 hours in the current international ongoing HI-DEF test. In theory, the earlier, the better curative effect. So this experiment is more likely to get a better curative effect. Xingnaojing injection is widely used in clinical in china, but lack of rigorous randomized controlled trial to prove its brain protection effect currently. Successful completion of this study will provide a crucial, reliable experimental evidence for a new treatment for acute cerebral hemorrhage. ICH is one of main causes of disability and death. A successful study demonstrating the efficacy of DFO and xingnaojing injection would be of considerable public health significance.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 80 years
2. The diagnosis of ICH is confirmed by brain CT scan
3. NIHSS score ≥ 6 and GCS > 6 upon presentation
4. The first dose of the study drug can be administered within 12h of ICH symptom onset
5. Functional independence prior to ICH, defined as pre-ICH mRS ≤ 1
6. Signed and dated informed consent is obtained.

Exclusion Criteria:

1. Known hypersensitivity to deferoxamine or xingnaojing injection
2. Known severe iron deficiency anemia (defined as hemoglobin concentration < 7g/dL or requiring blood transfusions)
3. Abnormal renal function, defined as serum creatinine > 2 mg/dL
4. Planned surgical evacuation of ICH prior to administration of study drug
5. Suspected secondary ICH related to tumour, ruptured aneurysm or arteriovenous malformation, hemorrhagic transformation of an ischemic infarct, or venous sinus thrombosis
6. Infratentorial hemorrhage
7. Irreversibly impaired brainstem function (bilateral fixed and dilated pupils and extensor motor posturing)
8. Complete unconsciousness, defined as a score of 3 on item 1a of the NIHSS (Responds only with reflex motor or autonomic effects or totally unresponsive, and flaccid)
9. Pre-existing disability, defined as pre-ICH mRS ≥ 2
10. Coagulopathy - defined as elevated aPTT or INR >1.3 upon presentation; concurrent use of direct thrombin inhibitors (such as dabigatran), direct factor Xa inhibitors (such as rivaroxaban), or low-molecular-weight heparin
11. Taking iron supplements containing ≥ 325 mg of ferrous iron
12. Patients with heart failure taking > 500 mg of vitamin C daily
13. Known severe hearing loss
14. Known pregnancy, or positive pregnancy test, or breastfeeding
15. Patients known or suspected of not being able to comply with the study protocol due to alcoholism, drug dependency, noncompliance, living in another state or any other cause
16. Life expectancy of less than 90 days due to comorbid conditions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Numbers of patients with the perihematomal edema (PHE) volume variation. | 7 days
  decreases of more than 20% from initial PHE volumes were defined as "decreased" PHE volume; increases of more than 20% from initial PHE volumes were defined as "increased" PHE volume; changes between -20% and 20% were defined as "unchanged".

SECONDARY OUTCOMES:
The residual cavity volume | 90 days
  the variation of residual cavity volume of
The variation of the mRS score and the Bathel Index | 90 days
  the variation of mRS score and Bathel Index of different treated subjects from ICH onset to treatment time windows.
mortality | 90 days
  the mortality of different treated subjects from ICH onset to treatment time windows.
Frequency of Treatment-related Adverse Events | 90 days
  The safety endpoints will include all DFO-related adverse events until day-7 or discharge (whichever is earlier), and DFO-related SAEs and through day-90.

CONTACTS AND LOCATIONS:
Overall Officials: Maolin He, MD, Principal Investigator — Department of Neurology，Beijing Shijitan Hospital，Capital Medical University
Locations (1):
- Department of Neurology，Beijing Shijitan Hospital，Capital Medical University, Beijing, China

REFERENCES:
- [Background] Okauchi M, Hua Y, Keep RF, Morgenstern LB, Schallert T, Xi G. Deferoxamine treatment for intracerebral hemorrhage in aged rats: therapeutic time window and optimal duration. Stroke. 2010 Feb;41(2):375-82. doi: 10.1161/STROKEAHA.109.569830. Epub 2009 Dec 31. PMID 20044521
- [Background] Selim M. Deferoxamine mesylate: a new hope for intracerebral hemorrhage: from bench to clinical trials. Stroke. 2009 Mar;40(3 Suppl):S90-1. doi: 10.1161/STROKEAHA.108.533125. Epub 2008 Dec 8. PMID 19064798
- [Background] Selim M, Yeatts S, Goldstein JN, Gomes J, Greenberg S, Morgenstern LB, Schlaug G, Torbey M, Waldman B, Xi G, Palesch Y; Deferoxamine Mesylate in Intracerebral Hemorrhage Investigators. Safety and tolerability of deferoxamine mesylate in patients with acute intracerebral hemorrhage. Stroke. 2011 Nov;42(11):3067-74. doi: 10.1161/STROKEAHA.111.617589. Epub 2011 Aug 25. PMID 21868742
- [Background] Morgenstern LB, Hemphill JC 3rd, Anderson C, Becker K, Broderick JP, Connolly ES Jr, Greenberg SM, Huang JN, MacDonald RL, Messe SR, Mitchell PH, Selim M, Tamargo RJ; American Heart Association Stroke Council and Council on Cardiovascular Nursing. Guidelines for the management of spontaneous intracerebral hemorrhage: a guideline for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2010 Sep;41(9):2108-29. doi: 10.1161/STR.0b013e3181ec611b. Epub 2010 Jul 22. PMID 20651276
- [Background] Chaudhary N, Gemmete JJ, Thompson BG, Xi G, Pandey AS. Iron--potential therapeutic target in hemorrhagic stroke. World Neurosurg. 2013 Jan;79(1):7-9. doi: 10.1016/j.wneu.2012.11.048. Epub 2012 Nov 19. No abstract available. PMID 23174156
- [Background] Demchuk AM, Dowlatshahi D, Rodriguez-Luna D, Molina CA, Blas YS, Dzialowski I, Kobayashi A, Boulanger JM, Lum C, Gubitz G, Padma V, Roy J, Kase CS, Kosior J, Bhatia R, Tymchuk S, Subramaniam S, Gladstone DJ, Hill MD, Aviv RI; PREDICT/Sunnybrook ICH CTA study group. Prediction of haematoma growth and outcome in patients with intracerebral haemorrhage using the CT-angiography spot sign (PREDICT): a prospective observational study. Lancet Neurol. 2012 Apr;11(4):307-14. doi: 10.1016/S1474-4422(12)70038-8. Epub 2012 Mar 8. PMID 22405630
- [Background] Gu Y, Hua Y, Keep RF, Morgenstern LB, Xi G. Deferoxamine reduces intracerebral hematoma-induced iron accumulation and neuronal death in piglets. Stroke. 2009 Jun;40(6):2241-3. doi: 10.1161/STROKEAHA.108.539536. Epub 2009 Apr 16. PMID 19372448
- [Background] Okauchi M, Hua Y, Keep RF, Morgenstern LB, Xi G. Effects of deferoxamine on intracerebral hemorrhage-induced brain injury in aged rats. Stroke. 2009 May;40(5):1858-63. doi: 10.1161/STROKEAHA.108.535765. Epub 2009 Mar 12. PMID 19286595